CLINICAL TRIAL: NCT05802069
Title: Medical College of Wisconsin Master Predict (Profile Related Evidence Determining Individualized Cancer)
Brief Title: MCW Master Predict (Profile Related Evidence Determining Individualized Cancer Therapy)
Status: Recruiting | Type: Observational
Sponsor: Sameem M. Abedin, MD (Other)
Responsible Party: Sponsor-Investigator, Sameem M. Abedin, MD, Assistant Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: PRO00044894
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A primary objective is to enable prospective collection of blood, urine, and other tissues for the purpose of identifying markers of outcomes, including, but not limited to genomic, immunologic, and pharmacologic profile testing from patients with cancer and related disorders at MCW/FH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is an observational trial for patients undergoing cancer-related interventions and therapy at Medical College of Wisconsin Cancer Center. Projects under this protocol will use patient data that will be collected both retrospectively and prospectively. It will also enable prospective sample collection for specific cancer-related studies.

DETAILED DESCRIPTION:
This is a master protocol that enables investigators to conduct observational research and correlative biospecimen studies. This study is non-therapeutic, with retrospective and prospective components. This will be a single-site study at MCW/FH. Retrospective data and, with consent, prospective observational data will be collected. The study will also include an opportunity for patients to consent to the analysis of specimens collected prospectively during care and for the collection of research-related testing of blood, stool, and/or urine. It is designed to decrease the burden on both patients and investigators by allowing consent to a protocol that will enable multiple minimal-risk studies.

Studies under this master protocol may perform data analysis using standard statistical techniques, as well as with advanced bioinformatics, machine learning, artificial intelligence, and other related technologies.

Collection and testing of biospecimens will only be performed if a proposed study that falls under this master protocol requires it. Studies may include a variety of simple or advanced techniques related to chemical, hematologic, molecular, proteomic, transcriptomic, immunomic, and metabolic analyses, as well as related multi-omic analysis for biomarker discovery, understanding correlations between treatment and molecular features, and/or for pharmacokinetic (PK) and pharmacodynamic (PD) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and older who were previously or are currently receiving care for a cancer-related condition at MCW/FH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who were previously or are currently receiving care for a cancer-related condition at MCW/FH. Newly diagnosed cancer patients at MCW/FH will also be considered. Patients must be willing and able to give informed consent for any prospective data or specimen collection.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects receiving precision therapies providing biospecimens of any kind. | One year
  Precision therapies are targeted against specific genomic mutations.
Number of subjects not receiving precision therapies and providing biospecimens. | One year
  Precision therapies are targeted against specific genomic mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Sameem Abedin, MD, Principal Investigator — Medical College of Wisconsin; Razelle Kurzrock, MD, Principal Investigator — Medical College of Wisconsin; Mary M. Horowitz, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No